CLINICAL TRIAL: NCT01241747
Title: Exercise for Women With Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma Center for the Advancement of Science and Technology (Other); Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR09-035
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Peripheral Artery Disease; Claudication; Women
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervised Exercise (Experimental): Supervised program consisting of graded treadmill walking, with progressive increments in exercise duration from 15 to 40 minutes at an exercise intensity of 40% of exercise capacity.
  Interventions: Behavioral: Walking Exercise
- Control (Active Comparator): Light resistance training without any walking
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Walking Exercise — 3 times per week for 3 months
  Arms: Supervised Exercise
Behavioral: Control — Resistance training 3 times per week for 3 months
  Arms: Control

SUMMARY:
Hypothesis #1. Supervised exercise rehabilitation will result in greater increases in exercise performance, peripheral vascular function, and health-related quality of life than compared to the attention-control group.

Hypothesis #2. The change in peripheral vascular function will be predictive of improved exercise performance following the supervised exercise program.

ELIGIBILITY:
Inclusion Criteria:

* women 60 years of age and older having a positive history of intermittent claudication assessed by the San Diego Claudication Questionnaire
* exercise limited by intermittent claudication during a screening treadmill test using the Gardner protocol
* an ankle/brachial index (ABI) < 0.90 at rest or < 0.73 immediately following the treadmill exercise test
* at least one year past menopause

Exclusion Criteria:

* absence of PAD (peripheral artery disease)
* asymptomatic PAD (Fontaine stage I)
* rest pain due to PAD (Fontaine stage III)
* tissue loss due to PAD (Fontaine stage IV)
* medical conditions that are contraindicative for exercise according to the American College of Sports Medicine (e.g., acute myocardial infarction, unstable angina, etc.)
* use of medications indicated for the treatment of intermittent claudication (cilostazol and pentoxifylline) initiated within three months prior to investigation)
* cognitive dysfunction (mini-mental state examination score < 24)
* active cancer, renal disease, or liver disease
* a calf skin fold measurement > 50 mm, because of potential interference with the light path of the near-infrared spectroscopy probe from penetrating the subcutaneous tissue
* pulse arterial oxygen saturation of the index finger < 95% because of the potential deleterious effect on calf muscle StO2 from poor pulmonary gas exchange

Ages: 60 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in walking distance to onset of leg pain and the change in walking distance to maximal leg pain | 3 months
Change in 6-minute walk distance | 3 months

SECONDARY OUTCOMES:
Change in calf muscle oxygen saturation | 3 months
Change in daily ambulatory activity | 3 months
Change in walking economy | 3 months
Change in peak oxygen uptake | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Gardner, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Clinical Research Center, Penn State College of Medicine, Hershey, Pennsylvania, United States

REFERENCES:
- [Result] Gardner AW, Poehlman ET. Exercise rehabilitation programs for the treatment of claudication pain. A meta-analysis. JAMA. 1995 Sep 27;274(12):975-80. PMID 7674529
- [Result] Gardner AW, Katzel LI, Sorkin JD, Bradham DD, Hochberg MC, Flinn WR, Goldberg AP. Exercise rehabilitation improves functional outcomes and peripheral circulation in patients with intermittent claudication: a randomized controlled trial. J Am Geriatr Soc. 2001 Jun;49(6):755-62. doi: 10.1046/j.1532-5415.2001.49152.x. PMID 11454114
- [Result] Gardner AW, Katzel LI, Sorkin JD, Goldberg AP. Effects of long-term exercise rehabilitation on claudication distances in patients with peripheral arterial disease: a randomized controlled trial. J Cardiopulm Rehabil. 2002 May-Jun;22(3):192-8. doi: 10.1097/00008483-200205000-00011. PMID 12042688
- [Result] Gardner AW, Killewich LA, Montgomery PS, Katzel LI. Response to exercise rehabilitation in smoking and nonsmoking patients with intermittent claudication. J Vasc Surg. 2004 Mar;39(3):531-8. doi: 10.1016/j.jvs.2003.08.037. PMID 14981444
- [Result] Gardner AW, Montgomery PS, Flinn WR, Katzel LI. The effect of exercise intensity on the response to exercise rehabilitation in patients with intermittent claudication. J Vasc Surg. 2005 Oct;42(4):702-9. doi: 10.1016/j.jvs.2005.05.049. PMID 16242558